CLINICAL TRIAL: NCT02396446
Title: AbStats at the Bedside: Improving Patient Feeding Decisions Using an Abdominal Acoustic Score
Status: Withdrawn | Type: Observational
Why Stopped: This study was never completed because the company was not able to support the trial with devices.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Brennan Spiegel, Director of Health Services Research, Cedars-Sinai Medical Center
Other Study IDs: Pro00039256
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Fasting; Diet; Biosensing Techniques
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intervention group: Inpatients at CSMC whose abdominal acoustic sounds will be measured using the AbStats device.
  Interventions: Other: Abdominal acoustic measurement

INTERVENTIONS:
Other: Abdominal acoustic measurement — Device meant to listen to the sounds of the gut to determine post op ileus.

SUMMARY:
This study is being conducted to determine whether providers who have access to their patients' acoustic intestinal rate score as calculated by an abdominal acoustic sensor that continuously monitors bowel sounds (AbStats) will be more likely to advance their patients' diets to a solid diet sooner than those who do not have access to this rate. AbStats calculates intestinal rates by using two small sensors placed on a patient's abdomen to measure and analyze their abdominal sounds.

Patients will be asked to wear a sensor every morning for 20 minutes while they are fasting daily during their inpatient visit. The sensor will measure the sounds within their abdomen. This data will be interpreted by the AbStats device, which will provide an intestinal rate measurement based on the sounds recorded by the sensors.

This intestinal rate will be provided to the patient's treating physician together with other vital signs. The doctor, at his/her discretion, may choose to use this information to make decisions about the patient's feeding status.

DETAILED DESCRIPTION:
The research team will use an abdominal acoustic sensor that continuously monitors bowel sounds (AbStats) to obtain acoustic measurements from 50 Cedars-Sinai Medical Center (CSMC) hospital patients by placing a disposable sensor on their abdomen. The sensor will be connected to a bedside monitor which records the sounds collected by the sensors and interprets them to create an intestinal rate reading, measured as acoustic events per minute. The research team will enter this score into the patient's chart and make it available to the patient's clinician(s), to use at their discretion to make decisions on whether or not to advance their patient's diet based on intestinal rate interpretation guidelines previously developed. The entry will provide a numerical intestinal rate with a brief interpretation of the score as listed below. This will be based on interpretations of the measures provided by the AbStats bedside computer, which have been previously developed in a wider research study.6 The scores will be interpreted using the following criteria:

Fasting intestinal rate score of <3 per minute: Ileus; Consider holding diet advancement until there is more evidence of GI function (feeding "red light")

Fasting intestinal rate score of 3-5 per minute: Slow motility; Consider advancing to liquid diet if NPO, assuming it is otherwise medically and surgically appropriate (feeding "yellow light")

Fasting intestinal rate score of >5 per minute: Normal motility; consider advancing to full diet if medically and surgically appropriate (feeding "green light")

Even though these readings will be provided in the patient chart, physicians must use their clinical judgment and account for mental status, aspiration risk, medications, surgical and medical comorbidities before making any feeding decisions. The intestinal rate is merely a new piece of information that provides objective evidence of GI function; it is likely superior to current best practices, which are notoriously unreliable for truly determining GI functional status and motility.

The research team will discuss the project with the patient's medical teaching attending physician, and will request their approval prior to approaching a patient. Once the doctor's approval is secured, researchers will approach the patient and provide them with detailed information about the project activities. If they agree to participate, the AbStats sensor will be placed on the patient's abdomen every morning for 20 minutes while the patient is fasting for the duration of their hospital stay. The sensor will be connected to a bedside computer that will process the data and calculate an intestinal rate, which will appear on the AbStats' gateway screen. The rate and its time-stamp will be entered into the patient's CS-Link (CSMC's EHR) chart by the research team. Once the patient is discharged, their participation in the study will be completed.

After discharge, the patient's chart will be reviewed by a member of the research staff. Using the "Dietary Orders" section of the "Active Orders" tab of the "Patient Summary" section of the patients CS-Link chart, we will determine the length of time from fasting (NPO) to full diet for each patient, as X1-X0, where X1 is time of order to full diet and X0 is time of hospital admission as noted in the "Encounters" section of the patient chart. Full diet will be determined from a dietary order in the chart stating "Diet Regular". The time to full diet will be reported in hours.

Medical residents and members of the Cedars-Sinai Department of Health Services Research staff will collect the following data (measures) at the patient's bedside:

Patient time (hours) to advancement to solid diet Abdominal intestinal rate measured by AbStats disposable biosensor

ELIGIBILITY:
Inclusion Criteria:

* Awake and alert
* Not on a regular diet
* No mild to moderate acute pancreatitis
* No obstructed bowel not amenable to feeding tube placement beyond the obstruction
* No massive GI hemorrhage
* No impending or established toxic megacolon
* No colonic perforation
* No severe dysmotility making enteral feeding not possible
* No high output intestinal fistula
* Able to access the gut for enteral feeding
* No abdominal compartment syndrome
* No withdrawal of care/DNAR status
* No evidence of severe or prolonged ileus
* No hemodynamic compromise (MAP <60) requiring high dose vasopressors alone or in combination with large volume fluid or blood product resuscitation to maintain cellular perfusion
* No diffuse peritonitis
* No intractable vomiting
* Not pregnant
* At least 18 years of age

Exclusion Criteria:

* Not awake and alert
* On regular diet
* Mild to moderate acute pancreatitis
* Obstructed bowel not amenable to feeding tube placement beyond the obstruction
* Massive GI hemorrhage
* Impending or established toxic megacolon
* Bowel perforation
* Severe dysmotility making enteral feeding impossible
* High output intestinal fistula
* Unable to access the gut for enteral feeding
* Abdominal compartment syndrome
* Withdrawal of care/DNAR status
* Severe ileus with NG output >1200 ml/d or gastric residual volumes >400 with additional signs of intolerance including absence of bowel sounds, abdominal distention, presence of air/fluid levels on abdominal radiographs
* Hemodynamic compromise (MAP <60) requiring high dose vasopressors alone or in combination with large volume fluid or blood product resuscitation to maintain cellular perfusion
* Diffuse peritonitis
* Intractable vomiting
* Pregnant women
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients at CSMC
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of acoustic events | One minute
  Number of acoustic events recorded by the AbStats device in one minute.
Mean time to advancement to full diet | Inpatient visit
  Mean time to advance a patient to a full diet

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center

REFERENCES:
- [Background] Agarwal E, Ferguson M, Banks M, Batterham M, Bauer J, Capra S, Isenring E. Nutrition care practices in hospital wards: results from the Nutrition Care Day Survey 2010. Clin Nutr. 2012 Dec;31(6):995-1001. doi: 10.1016/j.clnu.2012.05.014. Epub 2012 Jun 18. PMID 22717261
- [Background] Barr J, Hecht M, Flavin KE, Khorana A, Gould MK. Outcomes in critically ill patients before and after the implementation of an evidence-based nutritional management protocol. Chest. 2004 Apr;125(4):1446-57. doi: 10.1378/chest.125.4.1446. PMID 15078758
- [Background] Villet S, Chiolero RL, Bollmann MD, Revelly JP, Cayeux R N MC, Delarue J, Berger MM. Negative impact of hypocaloric feeding and energy balance on clinical outcome in ICU patients. Clin Nutr. 2005 Aug;24(4):502-9. doi: 10.1016/j.clnu.2005.03.006. PMID 15899538
- [Background] Franklin GA, McClave SA, Hurt RT, Lowen CC, Stout AE, Stogner LL, Priest NL, Haffner ME, Deibel KR, Bose DL, Blandford BS, Hermann T, Anderson ME. Physician-delivered malnutrition: why do patients receive nothing by mouth or a clear liquid diet in a university hospital setting? JPEN J Parenter Enteral Nutr. 2011 May;35(3):337-42. doi: 10.1177/0148607110374060. Epub 2011 Mar 7. PMID 21383319
- [Background] McClave SA, Martindale RG, Vanek VW, McCarthy M, Roberts P, Taylor B, Ochoa JB, Napolitano L, Cresci G; A.S.P.E.N. Board of Directors; American College of Critical Care Medicine; Society of Critical Care Medicine. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):277-316. doi: 10.1177/0148607109335234. No abstract available. PMID 19398613
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837